CLINICAL TRIAL: NCT00504790
Title: A Phase I, Open-Label, Dose-Escalation, First Time in Human Study to Evaluate the Safety Profile, Pharmacokinetics, and Pharmacodynamics of GSK923295 in Subjects With Refractory Cancers
Brief Title: Phase I Study to Assess the Safety, Pharmacokinetics, & Pharmacodynamics of GSK923295 in Subjects w/ Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPE107602
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: GSK923295,; First Time in Human,; pharmacodynamics; cancer,; maximally tolerated dose, pharmacokinetics,; Refractory Cancer; CENPE,; Phase I,
MeSH Terms: conditions — Neoplasms | interventions — GSK923295

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK923295 (Experimental): anti-mitotic compound under study
  Interventions: Drug: GSK923295

INTERVENTIONS:
Drug: GSK923295 — anti-mitotic compound

SUMMARY:
This is a Phase I, open-label, first time in human study of GSK923295, in adult subjects with cancers that do not respond to standard therapy. This study will be conducted in two stages; a dose-escalation stage (Stage 1) and an expansion cohort stage (Stage 2).

DETAILED DESCRIPTION:
Centromere-associated protein E (CENP-E) is a protein that is required for correct chromosomal alignment in mitosis. Loss of CENP-E activity, due to microinjection of antibodies, ablation of gene expression with siRNA or antisense oligonucleotides, or inhibition of enzymatic activity by small molecule inhibitors, causes aberrant cell cycle arrest in mitosis, characterized by a bipolar mitotic spindle with misaligned chromosomes. Studies with small molecule inhibitors have demonstrated that this aberrant cell cycle arrest can result in apoptosis and cell death. CENP-E has been shown to be abundantly expressed in a variety of human tumors. GSK923295 is a potent and selective CENP-E inhibitor which has demonstrated potent and broad spectrum antitumor activity against solid and hematologic malignancies in vitro. GSK923295 is intended for use either as a monotherapy or in combination with existing anti-cancer therapies.

A drug targeting CENP-E may prove as efficacious as the taxanes and vinca alkaloids, without the potential for neurotoxicity or other side-effects associated with interference of tubulin function in non-dividing cells. Similar to many other anti-proliferative drugs, CENP-E inhibitors are expected to have manageable dose-limiting toxicities resulting from action on normal proliferating tissues (e.g., myelosuppression and gastrointestinal epithelial cell damage). The opportunity for inhibitors of CENP-E lies in the potential for broad efficacy. The absence of broad clinical experience with anti-mitotic cancer therapies acting on targets other than tubulin complicates prediction of additional benefits, beyond the lack of neurotoxicity that might accrue from a drug targeting CENPE.

The purpose of this Phase I, first time in human (FTIH) study in subjects with refractory cancers is to determine the maximally tolerated dose (MTD) (or recommended dose based on available safety, pharmacokinetic (PK) and response data), dose-limiting toxicities (DLTs), PK, pharmacodynamics (PD), and preliminary clinical activity of GSK923295, an inhibitor of CENP-E.

The primary objectives in Stage 1 (Dose Escalation) are:

• To determine the MTD (or recommended dose based on available safety, PK, and response data), DLTs, safety, and PK of GSK923295 administered to subjects with advanced, refractory malignancies.

The primary objectives in Stage 2 (Expansion Cohort) are:

• To evaluate the safety and PK of GSK923295 at the MTD (or recommended dose based on available safety, PK, and response data) administered to subjects with advanced, refractory malignancies.

Secondary Objectives in the study are:

* To determine the clinical activity of GSK923295 administered to subjects with advanced, refractory malignancies.
* To evaluate the effect of GSK923295 on biomarkers in normal host tissue (Stage 1 and 2) and tumor (Stage 2, optional in Stage 1) and the effect of GSK923295 on tumor metabolism with FDG-PET imaging (Stage 2, optional in Stage 1).
* Explore associations between biochemical and genetic characteristics of baseline archival tumor specimens (Stage 1 and Stage 2), biopsy-accessible tumor specimens (Stage 2), and anti-tumor response.
* Explore pharmacogenomic associations between genetic variants in drug metabolizing and drug transport genes and PK, safety, and efficacy of GSK923295.

The primary and secondary endpoint(s) used to assess the objective measures are:

Primary

• Adverse events (AE) and changes from baseline in vital signs, clinical laboratory parameters, and electrocardiography (ECG) assessments will be evaluated to assess safety profile.

Secondary

* The MTD (or recommended dose based on available safety, PK, and response data) where no more than 1 of 6 subjects has a DLT in the first treatment cycle.
* PK parameters CL, Vdss, AUC(0-∞), AUC(0-t), Cmax, tmax, and t1/2 (Stage 1) and develop a PK model for GSK923295 (Stage 1 and 2).
* Anti-tumor activity measurements will be obtained at baseline and after every second cycle according to the following:
* Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines for solid tumors (for solid tumors and non-Hodgkin's lymphoma).
* National Cancer Institute - Working Group (NCI-WG) Guidelines for chronic lymphocytic leukaemia.
* Exploratory PK/PD modeling of safety and response data.
* Changes in biomarkers of cell proliferation and cell death or imaging endpoints.
* Biomarker profiles in archival tumor specimens and their correlation with clinical activity.
* Genetic polymorphisms in key enzymes involved in the metabolism and disposition of GSK923295 and correlations with pharmacokinetic, safety, and response (pharmacodynamic) data.

The study will consist of two stages. Stage 1 consists of a dose escalation stage to determine the MTD (or recommended dose based on available safety, PK and response data) using an accelerated titration scheme combined with standard dose escalation methods. GSK923295 will be administered intravenously over one hour, once weekly for 3 consecutive weeks (i.e., Day 1, 8, and 15) with treatment cycles repeated every 4 weeks (each cycle = 28 days). During Stage 1, safety, pharmacokinetics, pharmacodynamics, and clinical activity will be assessed. Tumor biopsies and PET imaging are optional in Stage 1 subjects. The MTD (or recommended dose based on available safety, PK and response data) will be defined as the dose of GSK923295 at which no more than 1 of 6 subjects experiences a DLT in the first treatment cycle. Eighteen subjects are anticipated to participate in Stage 1 of the study. In Stage 2, 15-20 additional subjects will be enrolled at the MTD (or recommended dose based on available safety, PK and response data) dose to further evaluate the safety of GSK923295. In Stage 2, PK samples (using a sparse PK sampling scheme for population PK analyses), PET imaging, and tumor biopsies will be obtained. Clinical activity will be assessed. Subjects (Stage 1 and Stage 2) will remain on study until they meet the criteria for treatment discontinuation described in the protocol. It is anticipated that 33-38 subjects will participate in the study (18 in Stage 1 and 15-20 in Stage 2. During Stage 1 and Stage 2, subjects with histologically confirmed advanced refractory solid tumors will be enrolled. In Stage 2, subjects with refractory non-Hodgkin's lymphoma and chronic lymphocytic leukemia can also be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent provided.
* a) Stage 1 Subjects: Histologically or cytologically confirmed diagnosis of solid tumor malignancy that is not responsive to accepted standard therapies, or for which there is no standard therapy.

  b) Stage 2 Subjects: Histologically or cytologically confirmed diagnosis of solid tumor malignancy, non-Hodgkin's lymphoma, or chronic lymphocytic leukemia that is not responsive to accepted standard therapies, or for which there is no standard therapy.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* 18 years old or older.
* Male or female
* A female is eligible to enroll in the study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who:
  * Has had a hysterectomy, or
  * Has had a bilateral oophorectomy (ovariectomy), or
  * Has had a bilateral tubal ligation, or
  * Is post-menopausal (demonstrate total cessation of menses for greater than or equal to one year).
  * Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following from at least two weeks prior to study enrolment until completion of the Post Study procedures:
  * An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
  * Vasectomized partner who is sterile and is the sole sexual partner for that woman.
  * Complete abstinence from sexual intercourse.
  * Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; OR diaphragm with spermicide; OR male condom and diaphragm.
* A male is eligible to enter and participate in the study if he either agrees to abstain from sexual intercourse or use a condom and occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository from the first dose administered until completion of the Post-Treatment procedures; or is surgically sterile.
* Adequate organ systems function as defined in the protocol.
* Subjects may have measurable lesions according to RECIST criteria in Stage 1. It is required in Stage 2 that subjects with solid tumors have measurable lesions according to RECIST criteria.
* Paraffin-embedded archival tumor tissue available for testing.
* At least one target tumor accessible to serial core needle biopsies at study entry (screening) and one additional time point post-dose Cycle 1. Note: optional for Stage 1 (Dose Escalation); it is mandatory for Stage 2 (Expansion Cohort)

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Any major surgery OR prior anti-cancer therapy including but not limited to chemotherapy, radiotherapy, immunotherapy, biological therapy, or investigational therapy within the past 28 days (42 days for prior nitrosureas or mitomycin C).
* Prior allogeneic or autologous bone marrow transplant.
* Greater than 30% bone marrow irradiated.
* Unresolved toxicity ≥ Grade 2 from previous anti-cancer therapy (except alopecia).
* History of hemolytic anemia (either congenital or acquired) OR current laboratory evidence of hemolysis (Grade 1CTCAE or greater) that includes at least one of the following:

  * Decrease in serum haptoglobin (outside normal institutional laboratory values)
  * Increase in indirect bilirubin (outside normal institutional laboratory values)
  * Peripheral blood smear consistent with hemolysis (presence of schistocytes)
* Pre-existing peripheral neuropathy or other neurological toxicity ≥ Grade 2.
* Female subjects who are pregnant or lactating.
* Any serious or unstable pre-existing medical, psychiatric, active infection or other condition (including lab abnormalities) that could interfere with subject safety or obtaining informed consent.
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
* QTc prolongation defined as a QTc interval greater than or equal to 450 msecs.
* Other significant ECG abnormalities including 2nd or 3rd degree AV block or bradycardia (ventricular rate less than 50 beats/min).
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within the past 6 months.
* For subjects with a history of myocardial infarction, congestive heart failure, abnormal left ventricular ejection fraction (LVEF), or prior anthracycline exposure, LVEF must be assessed within 28 days of the first dose of study drug by one of the following methods: MUGA or ECHO. An LVEF measurement of < 50% will exclude the subject from participation in the study.
* Class III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Current use of warfarin ≥ 4 mg per day. NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted. PT/PTT must meet the inclusion criteria.
* Current use of prohibited medications in accordance with the guidelines detailed in the protocol in the "Prohibited Medications" section.
* Current use of drugs with risk of torsade de pointes as described in the protocol.
* Evidence of symptomatic or untreated central nervous system involvement (i.e., brain metastases, leptomeningeal disease, cord compression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-06-25 (Actual); Primary Completion 2012-05-07 (Actual); Study Completion 2012-05-08 (Actual)

PRIMARY OUTCOMES:
Safety: - physical exam | at screen & Day(D) 1 of each cycle and follow-up(F/U)
- vital signs and lab tests | at screen & D1, 8, 15, & 22 for each cycle & F/U
- ECGs | at screen and D1, 8 & 15 for each cycle & F/U
continuous monitoring of adverse events | each visit

SECONDARY OUTCOMES:
Plasma samples of GSK923295 taken at: | - Day 1 & 15 (Cycle 1) for Stage 1
  used to measure levels of the drug in blood over time
Plasma samples of GSK923295 taken at: | - Day 1 of each cycle for Stage 2
  used to monitor levels of the drug in blood

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Madison, Wisconsin

REFERENCES:
- [Result] Chung V, Fleming RA, Johnson BM, Gauvin J, Cyr TL, Lager JJ, Lu E, Alberti DB, Williams B, Weber BL, Synold T, Holen KD. A phase 1 and first time in human study of the centromere associated protein E (CENP-E) inhibitor GSK923295A in patients with advanced solid rumors. American Association of Clinical Research Annual Meeting 2008, Oral Presentation, Abstract LB 246
- [Result] Fleming RA, Holen KD, Cyr TL, Johnson BM, Gauvin JL, Lager JJ, Williams B, Alberti DB, Weber BL, Grilley-Olson JE, Chung V. A phase I dose escalation and pharmacokinetic study of the novel mitotic checkpoint inhibitor GSK923295A in patients with solid tumors. (Poster). EORTC/NCI/AACR Molecular Targets and Cancer Therapeutics Meeting, Geneva, Switzerland, 2008
- [Result] Holen KD, Heath E, Shelman WS, Kirby LC, Johnson BM, Botbyl JD, Grilley-Olson JE, Lampkin TA, Chung V. Phase I, first-in-human study of the centromere-associated protein e (CENP-E) inhibitor GSK923295 in patients with advanced solid tumors (Study CPE107602). American Society of Clinical Oncology 2010, Oral Presentation, Abstract 3012
- See also: Results for study CPE107602 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CPE107602?search=study&search_terms=CPE107602#rs